CLINICAL TRIAL: NCT00268086
Title: Constrictive Pericarditis in the Adult Congenital Cardiac Population
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-123
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Congenital Disorders
Keywords: constrictive pericarditis; adult congenital patients; pulmonary insufficiency
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Pericarditis, Constrictive; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The primary aim of this study is to determine the clinical and radiographic findings with constrictive pericarditis in the adult congenital population and determine the degree of right heart failure and dilation from pulmonary insufficiency in the presence of constrictive pericarditis

The secondary aim is to elucidate ways to better diagnose constrictive pericarditis and elucidate ways to diagnose right heart failure in the presence of constrictive pericarditis.

DETAILED DESCRIPTION:
Constrictive pericarditis is a notoriously difficult diagnosis to reach. There are no signs, symptoms or pathognomonic diagnostic tests for pericardial constriction. In the adult congenital patients, it is also difficult. In addition, with pulmonary insufficiency, constrictive pericarditis may mask the findings of progressive right sided ventricular dilation and heart failure.

The primary aim of this study is to determine the clinical and radiographic findings with constrictive pericarditis in the adult congenital population and determine the degree of right heart failure and dilation from pulmonary insufficiency in the presence of constrictive pericarditis

The secondary aim is to elucidate ways to better diagnose constrictive pericarditis and elucidate ways to diagnose right heart failure in the presence of constrictive pericarditis.

Study Design and Methodology:

Retrospective chart review - approximately 15 patients

Preoperative data:

ECHO and cath findings

Operative data:

Operative findings

Postoperative data:

ECHO and cath findings

ELIGIBILITY:
Inclusion Criteria:

* patients in the adult congenital heart disease clinic who have been diagnosed or operated on with constrictive pericarditis

Exclusion Criteria:

* those who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Kogon, MD, Principal Investigator — Emory Univ. SOM Cardiothoracic Surgery at Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States